CLINICAL TRIAL: NCT06975397
Title: The Effect of Kinesio Taping on Reducing Diastasis Recti Abdominis Size in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Proskura Patrycja (Other)
Responsible Party: Sponsor-Investigator, Proskura Patrycja, dr, Wroclaw University of Health and Sport Sciences
Organization: Wroclaw University of Health and Sport Sciences (Other)
Allocation: Not Applicable | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: No. 34/2018
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Diastasis Recti Abdominis (DRA)
Keywords: Diastasis recti abdominis; Kinesio Taping; Postpartum; Ultrasonography; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Who Masked: Participant
Masking Description: None of the participants were aware of group allocations or the interventions used in each group according to CONSORT's diagram. Each subject was given the same exercises (instructor-led) and tested individually to maintain study blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - no taping - control group (Sham Comparator): The eligibility criteria for the study were:
  * aged between 25 and 45 years
  * first singleton pregnancy
  * natural childbirth
  * no medical contraindications for exercising and taping.
  The exclusion criteria were:
  * childbirth through cesarean section
  * more than eight weeks from natural childbirth
  * body mass index (BMI) over 35 kg/m2
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Group 2 - taping without tension - placebo group (Sham Comparator): The eligibility criteria for the study were:
  * aged between 25 and 45 years
  * first singleton pregnancy
  * natural childbirth
  * no medical contraindications for exercising and taping.
  The exclusion criteria were:
  * childbirth through cesarean section
  * more than eight weeks from natural childbirth
  * body mass index (BMI) over 35 kg/m2
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION; Other: kinesio taping
- Group 3 - taping at 50 % tension - tape group (Active Comparator): The eligibility criteria for the study were:
  * aged between 25 and 45 years
  * first singleton pregnancy
  * natural childbirth
  * no medical contraindications for exercising and taping.
  The exclusion criteria were:
  * childbirth through cesarean section
  * more than eight weeks from natural childbirth
  * body mass index (BMI) over 35 kg/m2
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION; Other: kinesio taping

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — This training and research project was conducted over eight weeks and started 6 - 8 weeks after natural childbirth. All study participants were included in the exercise program designed for postpartum females. Exercises included four sets that changed every two weeks and were held individually with a physiotherapist three times a week, every two to three days, for 45 minutes each unit. All participants performed breathing exercises, body posture correction, abdominal muscle strengthening exercises (transverse, oblique, and rectus abdominis muscles), and engaged other muscles to improve overall physical fitness.
Other: kinesio taping — The Kinesiology Tape used in this study has a European quality certificate (CE). Before the exercise program, on the day of the first ultrasound, participants had tapes placed on their abdomens. The tape length for each participant was 20 cm to ensure the ends were located on the lateral edges of the rectus abdominis muscles. Both ends of the tape were simultaneously attached to the abdomen, with two attached from the navel line upwards and one below it Each participant in the tape group was asked to breathe in using the abdominal muscles, and after a maximal stretch of the abdominal integuments, three tapes were attached at 50% tension or without tension. The taping procedure was repeated once per week, with the tapes attached for six days and removed at the end of the 6th day. The placebo and tape groups had a break on the 7th day
  Arms: Group 2 - taping without tension - placebo group; Group 3 - taping at 50 % tension - tape group

SUMMARY:
A three-arm parallel-group randomized controlled trial was conducted with 90 women aged 23-42 years, 6-8 weeks postpartum. Participants were randomly assigned to one of three groups: no kinesiotaping (control), placebo kinesiotaping (no tension), and kinesiotaping with 50% tension. All participants followed the same exercise program. The primary outcome measure was the Diastasis Recti Index (DRI), assessed via ultrasound at baseline, 4 weeks, and 8 weeks.

DETAILED DESCRIPTION:
This was a three-arm, parallel-group, randomised controlled trial with concealed allocation. The allocation of subjects to the experiment was arranged chronologically. Each woman meeting the inclusion criteria was consecutively qualified. None of the participants were aware of group allocations or the interventions used in each group according to CONSORT's diagram. Each subject was given the same exercises (instructor-led) and tested individually to maintain study blinding.

The clinical rationale for reducing DRA using Kinesio taping was evaluated in 90 females in the late postpartum period, defined as 6 - 8 weeks after childbirth.

The eligibility criteria for the study were:

* aged between 25 and 45 years
* first singleton pregnancy
* natural childbirth
* no medical contraindications for exercising and taping.

The exclusion criteria were:

* childbirth through cesarean section
* more than eight weeks from natural childbirth
* body mass index (BMI) over 35 kg/m2

All study participants were randomly divided into three groups of 30:

* Group 1 - no taping - control group,
* Group 2 - taping without tension - placebo group,
* Group 3 - taping at 50 % tension - tape group. There were no statistically significant differences in body dimensions between the study groups. All participants followed the same exercise program designed for postpartum females (Additional material - presentation of the exercise program). A Tanita electronic scale measured body weight and height. Examinations were conducted once per session at the beginning of the project and in the 4th and 8th weeks of training. Ultrasound examination used the Mindray DP10 apparatus (38 mm linear transducer) at a frequency of 5.0, 7.5, and 10.0 MHz and was performed by an ultrasound-trained physiotherapist. Two points were marked in a straight line with the cursor, the right and the left medial edge of the rectus muscle, and the inter-rectus distance was measured with an accuracy of 0.2 cm. Measurements were recorded at the navel line, 4.5 cm above, and 4.5 cm under the navel. Also, waist circumference measurement used a tailor's tape (with 0.2 cm accuracy), which was measured midway between the edge of the tenth rib and the highest point of the iliac crest. Inter-rectus distance and waist circumference were measured by the same person (the first author of the paper) over three project sessions. The DRA width at the given measurement line was normalized by waist circumference taken during the same measurement, which allowed the DRA width to be independently comparable to each subject's body dimensions.

This training and research project was conducted over eight weeks and started 6 - 8 weeks after natural childbirth. All study participants were included in the exercise program designed for postpartum females. Exercises included four sets that changed every two weeks and were held individually with a physiotherapist three times a week, every two to three days, for 45 minutes each unit. All participants performed breathing exercises, body posture correction, abdominal muscle strengthening exercises (transverse, oblique, and rectus abdominis muscles), and engaged other muscles to improve overall physical fitness.

The Kinesiology Tape used in this study has a European quality certificate (CE). Before the exercise program, on the day of the first ultrasound, participants had tapes placed on their abdomens. The tape length for each participant was 20 cm to ensure the ends were located on the lateral edges of the rectus abdominis muscles. Both ends of the tape were simultaneously attached to the abdomen, with two attached from the navel line upwards and one below it.

Each participant in the tape group was asked to breathe in using the abdominal muscles, and after a maximal stretch of the abdominal integuments, three tapes were attached at 50% tension or without tension. The detailed procedure for applying Kinesiology tape is described in Additional material. The taping procedure was repeated once per week, with the tapes attached for six days and removed at the end of the 6th day. The placebo and tape groups had a break on the 7th day, and the scheme was repeated for 8 weeks. After 4 weeks, a second ultrasound similar to the first measurement of the rectus abdominis muscle was performed as before. The 3rd measurement was taken after completing the exercise program, which took 8 weeks. Primary outcome: Diastasis Recti Index (DRI) was computed in order to normalize the ultrasound examination results. The DRA width was divided by waist circumference and multiplied by 100% to determine the changes in diastasis width at the navel line (DRIn), above the navel (DRIan), and under the navel (DRIun): DRI [%]=DRAw[cm]/(waist circumference [cm] )*100% where

* DRAw is the diastasis recti abdominis width at a given measurement line: at the navel, above the navel, and under the navel (respectively)
* waist circumference was measured at the navel line in a given session. The DRI index expressed as a percentage of waist circumference makes it possible to compare diastasis width changes dependently of body size. A zero DRI value does not mean that the linea alba is zero width. Normal linea alba at the navel line is approximately 2.24 cm ± 0.8 cm. A higher DRI points to a worse therapy outcome, and a DRI decrease indicates an improved result. The best result of DRI = 0 represents normal linea alba width and no DRA.

The effectiveness of Kinesio taping was assessed based on intergroup differences in the initial

measurement values (DRI1) taken before the start of the project, the second measurement after 4 weeks (DRI2), and the third measurement after 8 weeks (DRI3). The intergroup analysis compared the measurements taken at the navel line, above the navel, and under the navel. Determining the significance of intergroup differences between the three subsequent DRI scores will make it possible to determine the optimal therapy duration for obtaining the desired effects. Meanwhile, intragroup changes in the DRI reflect the effect of a given treatment, including exercise alone, exercise in combination with taping without tension, and exercise with taping at 50% tension.

ELIGIBILITY:
Inclusion Criteria:

* - aged between 25 and 45 years
* first singleton pregnancy
* natural childbirth
* no medical contraindications for exercising and taping.

Exclusion Criteria:

* - childbirth through cesarean section
* more than eight weeks from natural childbirth
* body mass index (BMI) over 35 kg/m2

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The eligibility criteria for the study were:
  * aged between 25 and 45 years
  * first singleton pregnancy
  * natural childbirth
  * no medical contraindications for exercising and taping.
  The exclusion criteria were:
  * childbirth through cesarean section
  * more than eight weeks from natural childbirth
  * body mass index (BMI) over 35 kg/m2
Enrollment: 161 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
Diastasis Recti Index (DRI) | The effectiveness of Kinesio taping was assessed based on intergroup differences in the initial measurement values (DRI1) taken before the start of the project, the second measurement after 4 weeks (DRI2), and the third measurement after 8 weeks (DRI3).
  outcome: Diastasis Recti Index (DRI) was computed in order to normalize the ultrasound examination results. The DRA width was divided by waist circumference and multiplied by 100% to determine the changes in diastasis width at the navel line (DRIn), above the navel (DRIan), and under the navel (DRIun): DRI [%]=DRAw[cm]/(waist circumference [cm] )*100% where
  * DRAw is the diastasis recti abdominis width at a given measurement line: at the navel, above the navel, and under the navel (respectively)
  * waist circumference was measured at the navel line in a given session.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kmieć-Nowakowska, PhD, Principal Investigator — Joanna Kmieć-Nowakowska Circa Feminae - terapia dla kobiet Ul. Abramowskiego 41 Wrocław nip 8981976347
Locations (1):
- Rehafit, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the lack of participant consent for data sharing and protect privacy in accordance with data protection regulations.

REFERENCES:
- [Background] Tuttle LJ, Fasching J, Keller A, Patel M, Saville C, Schlaff R, Walker A, Mason M, Gombatto SP 2018 Noninvasive Treatment of Postpartum Diastasis Recti Abdominis. Journal of Women's Health Physical Therapy 42(2): 65-75, doi:10.1097/jwh.0000000000000101
- [Background] Torbe D, Stolarek A, Lubkowska A, Torbe A. [Physical activity recommended in the early postpartum period]. Pomeranian J Life Sci. 2016;62(3):53-6. Polish. PMID 29537766
- [Background] Rath AM, Attali P, Dumas JL, Goldlust D, Zhang J, Chevrel JP. The abdominal linea alba: an anatomo-radiologic and biomechanical study. Surg Radiol Anat. 1996;18(4):281-8. doi: 10.1007/BF01627606. PMID 8983107
- [Background] Ptaszkowska L, Gorecka J, Paprocka-Borowicz M, Walewicz K, Jarzab S, Majewska-Pulsakowska M, Gorka-Dynysiewicz J, Jenczura A, Ptaszkowski K. Immediate Effects of Kinesio Taping on Rectus Abdominis Diastasis in Postpartum Women-Preliminary Report. J Clin Med. 2021 Oct 28;10(21):5043. doi: 10.3390/jcm10215043. PMID 34768563
- [Background] Pawar PA, Yeole UL, Navale M, Patil K 2020 Effect of kinesiotaping on diastasis recti in post-partum women. Indian Journal of Public Health Research & Development 11(6):689-94, https://doi.org/10.37506/ijphrd.v11i6.9865
- [Background] O'Sullivan D, Bird SP 2011 Utilization of Kinesio Taping for Fascia Unloading. International Journal of Athletic Therapy and Training 16(4): 21-27, https://doi.org/10.1123/ijatt.16.4.21
- [Background] Mullins E, Sharma S, McGregor AH. Postnatal exercise interventions: a systematic review of adherence and effect. BMJ Open. 2021 Sep 30;11(9):e044567. doi: 10.1136/bmjopen-2020-044567. PMID 34593482
- [Background] Mota P, Pascoal AG, Carita AI, Bo K. Normal width of the inter-recti distance in pregnant and postpartum primiparous women. Musculoskelet Sci Pract. 2018 Jun;35:34-37. doi: 10.1016/j.msksp.2018.02.004. Epub 2018 Feb 20. PMID 29494833
- [Background] Mosiejczuk H, Lubinska A, Ptak M, Szylinska A, Kemicer-Chmielewska E, Laszczynska M, Rotter I. [Kinesiotaping as an interdisciplinary therapeutic method]. Pomeranian J Life Sci. 2016;62(1):60-6. Polish. PMID 29533589
- [Background] Michalska A, Rokita W, Wolder D, Pogorzelska J, Kaczmarczyk K. Diastasis recti abdominis - a review of treatment methods. Ginekol Pol. 2018;89(2):97-101. doi: 10.5603/GP.a2018.0016. PMID 29512814
- [Background] Mędrak A, Król T, Michałek-Król K, Dąbrowska-Galas M 2017 Kinesiotaping and the placebo effect. Family Medicine 20(4): 304-309, doi: 10.25121/MR.2017.20.4.304
- [Background] Mak DN, Au IP, Chan M, Chan ZY, An WW, Zhang JH, Draper D, Cheung RT. Placebo effect of facilitatory Kinesio tape on muscle activity and muscle strength. Physiother Theory Pract. 2019 Feb;35(2):157-162. doi: 10.1080/09593985.2018.1441936. Epub 2018 Feb 20. PMID 29461139
- [Background] Mady MM 2018 Kinesiotaping Therapy Techniquesfor Treating Postpartum Rectus Diastases: A Comparative Study. IOSR Journal of Nursing and Health Science 7:67-74, doi: 10.9790/1959-0703026774
- [Background] Lim C, Park Y, Bae Y. The effect of the kinesio taping and spiral taping on menstrual pain and premenstrual syndrome. J Phys Ther Sci. 2013 Jul;25(7):761-4. doi: 10.1589/jpts.25.761. Epub 2013 Aug 20. PMID 24259847
- [Background] Lemoncito MV, Paz-Pacheco E, Lim-Abrahan MA, Jasul G, Isip-Tan T, Sison CM 2010 Impact of Waist Circumference Measurement Variation on the Diagnosis of Metabolic Syndrome. Philippine Journal of Internal Medicine 48(3): 7-12
- [Background] Kirk B, Elliott-Burke T. The effect of visceral manipulation on Diastasis Recti Abdominis (DRA): A case series. J Bodyw Mov Ther. 2021 Apr;26:471-480. doi: 10.1016/j.jbmt.2020.06.007. Epub 2020 Aug 6. PMID 33992284
- [Background] Kase K, Wallis J, Kase T 2013 Clinical Therapeutic Applications of the Kinesio Taping Method. Tokyo, Japan: Ken Ikai Co Ltd
- [Background] Keeler J, Albrecht M, Eberhardt LA, Horn L, Donnelly C, Lowe D 2012 Diastasis Recti Abdominis: A Survey of Women's Health Specialists for Current Physical Therapy Clinical Practice for Postpartum Women. Journal of Women's & Pelvic Health Physical Theray 36: 131-142, doi:10.1097/JWH.0B013E318276F35F
- [Background] Izydorczyk B, Walenista W, Kamionka A, Lizinczyk S, Ptak M. Connections Between Perceived Social Support and the Body Image in the Group of Women With Diastasis Recti Abdominis. Front Psychol. 2021 Aug 9;12:707775. doi: 10.3389/fpsyg.2021.707775. eCollection 2021. PMID 34434150
- [Background] Inge P, Orchard JJ, Purdue R, Orchard JW. Exercise after pregnancy. Aust J Gen Pract. 2022 Mar;51(3):117-121. doi: 10.31128/AJGP-09-21-6181. PMID 35224572
- [Background] Coldron Y, Stokes MJ, Newham DJ, Cook K. Postpartum characteristics of rectus abdominis on ultrasound imaging. Man Ther. 2008 May;13(2):112-21. doi: 10.1016/j.math.2006.10.001. Epub 2007 Jan 5. PMID 17208034
- [Background] Boissonnault JS, Blaschak MJ. Incidence of diastasis recti abdominis during the childbearing year. Phys Ther. 1988 Jul;68(7):1082-6. doi: 10.1093/ptj/68.7.1082. PMID 2968609
- [Background] Awad MA, Mahmoud AM, El-Ghazaly HM, Tawfeek RM 2017 Effect of Kinesio Taping on diastasis recti. Medical Journal Cairo University 85(6): 2289-2296
- [Background] Gluppe SB, Ellstrom Engh M, Bo K. Curl-up exercises improve abdominal muscle strength without worsening inter-recti distance in women with diastasis recti abdominis postpartum: a randomised controlled trial. J Physiother. 2023 Jul;69(3):160-167. doi: 10.1016/j.jphys.2023.05.017. Epub 2023 Jun 5. PMID 37286390
- [Background] Gilleard WL, Brown JM. Structure and function of the abdominal muscles in primigravid subjects during pregnancy and the immediate postbirth period. Phys Ther. 1996 Jul;76(7):750-62. doi: 10.1093/ptj/76.7.750. PMID 8677279
- [Background] Flament JB. [Functional anatomy of the abdominal wall]. Chirurg. 2006 May;77(5):401-7. doi: 10.1007/s00104-006-1184-5. German. PMID 16703394
- [Background] Fernandes da Mota PG, Pascoal AG, Carita AI, Bo K. Prevalence and risk factors of diastasis recti abdominis from late pregnancy to 6 months postpartum, and relationship with lumbo-pelvic pain. Man Ther. 2015 Feb;20(1):200-5. doi: 10.1016/j.math.2014.09.002. Epub 2014 Sep 19. PMID 25282439
- See also: WHO RECOMMENDATIONS — http://www.who.int/europe/news-room/fact-sheets/item/a-healthy-lifestyle---who-recommendations